CLINICAL TRIAL: NCT07076875
Title: Qualitative and Quantitative Assessment of Parental Satisfaction and Parental Care of Dental Care and Dental Services Provided in the Pediatric Dentistry Department in El Kasr El Einy: A Cross-sectional Study
Brief Title: Parental Satisfaction With Pediatric Dental Care at El Kasr El Einy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdullah Saad mohammed Alobaidan, M.D. Pediatric Dentistry, Cairo University
Other Study IDs: 10.11.23
Record Dates: First submitted 2025-05-29; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Dentistry; Health Services Accessibility; Patient Satisfaction; Dental Care for Children; Health Services Utilization
Keywords: Pediatric dental satisfaction; Dental access barriers Egypt; Parental dental experience; Unmet pediatric dental needs; Public dental hospital evaluation
MeSH Terms: conditions — Patient Satisfaction; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parents of the patient from age 2 to 12 years old
  Interventions: Other: Questioner interview

INTERVENTIONS:
Other: Questioner interview — The 2 questionnaires were translated from English to standard Arabic comprised of three sections, general information, including data and sociodemographic factors such as region of residence, parental education level, child age, child sex, and child order between siblings, Barriers to oral health care needs, including frequency and reasons for dental visits, any previous dental treatment, barriers to treatment such as fear of dentist, distance from the dental clinic, expense of an appointment due to health ban, responsibilities towards family members, not being familiar with appointment booking, and no available appointments, and Comprising of interviewer-administered questionnaires with a five-point Likert scale (strongly agree, agree, uncertain, disagree, strongly disagree) to assess the level of patients' satisfaction with the dental services provided.

SUMMARY:
This study aims to evaluate the barriers and unmet needs in utilizing dental services for children and measure parental satisfaction with the services provided at the Pediatric Department, Faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
This observational study evaluates barriers to dental service utilization, unmet treatment needs, and parental satisfaction within the Pediatric Dentistry Department at Cairo University's Faculty of Dentistry. All participants will complete a validated, interviewer-administered Arabic questionnaire assessing Sociodemographic factors (income, education, insurance), access barriers (financial, geographic, systemic, psychosocial via nineteen-item Likert scale), unmet dental needs (DMFT index, untreated conditions from electronic health records), parental satisfaction (nine-item scale evaluating service quality, staff attitudes, waiting times, and facilities). The study aims to generate evidence for optimizing pediatric dental care delivery in Egypt's largest academic dental center.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 2 to 12 years old

Exclusion Criteria:

* Parents refuse to sign the informed consent

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A group of parents who use dental services for their children that is from 2-12 years and attending faculty of dentistry pediatric department
Sampling Method: Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Parents' satisfaction | 6 months
  Evaluation of parents' satisfaction with the service provided in the dental clinic for their children by The structured and validated questionnaire consists of
  1. quantitative closed questions. The measurement unit includes both a nominal scale (%) and a quantitative scale (minutes).
  2. Qualitative open-ended questions. The measurement unit incorporates a nominal scale (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes